CLINICAL TRIAL: NCT02157285
Title: The Influence of Peer Mentoring on Contraceptive Decision Making Among Adolescents
Brief Title: Influence of Peer Mentoring on Adolescent Contraceptive Decision Making
Acronym: ImPACCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Courtney Schreiber, Director, Fellowship in Family Planning, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 816769
Record Dates: First submitted 2013-03-19; First posted 2014-06-05 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: Peer Counseling; LARC Desire
Keywords: Unintended pregnancy in adolescence; LARC; contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Routine Counseling (No Intervention): Subjects randomized to receive routine counseling before selecting a method of contraception
- Peer Mentor counseling (Experimental): Subjects randomized to receive peer counseling before selecting a method of contraception
  Interventions: Behavioral: Peer Mentor Counseling

INTERVENTIONS:
Behavioral: Peer Mentor Counseling — Peer mentoring will entail the peer mentor describing her positive experience with her LARC method. The participant will then have a chance to ask any experience related questions to the mentor. Any clinical inquiries or questions the mentor does not feel comfortable answering, she will defer to the contraceptive counselor/ physician who will be subsequently providing the routine counseling. The entire peer mentor encounter should not last more than 10 minutes.
  Arms: Peer Mentor counseling

SUMMARY:
This is a prospective, randomized-controlled trial in which subjects will be randomized to receive either routine contraceptive counseling or peer mentoring plus routine contraceptive counseling.

DETAILED DESCRIPTION:
Unintended adolescent pregnancy continues to be a significant public health problem in the United States. While the use of highly effective forms of birth control, such as the long-acting, reversible contraceptives (LARC) have been found to be more effective in decreasing pregnancy rates than non-LARC methods of birth control, knowledge and use of LARC has been shown to be low in this vulnerable population. We are interested in better understanding the influence peers may have on contraceptive decision making among adolescents. The purpose of this study is to evaluate the impact of a peer mentoring intervention on adolescent contraceptive decision making, specifically with regard to increasing long-acting, reversible contraceptive uptake. The main study intervention will consist of randomization to usual contraceptive counseling versus peer-mentoring plus usual contraceptive counseling. Pre- and post-intervention questionnaires will be used to better understand peer influence on contraceptive decision making, and to assess the peer mentor-teen intervention interaction.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Female
* Age 13-21 years old at enrollment
* Desiring contraception; either currently not taking any method of contraception, or not satisfied with current method, and not desiring pregnancy in the next 12 months
* Willing and able to follow the study protocol

Exclusion Criteria:

* Male gender
* Younger than 13 years old, older than 21 years old
* Pregnant or desiring pregnancy within the coming year
* Issues or concerns in the judgement of the investigator that may compromise the safety of the subject or confound the reliability of compliance and information acquired in this study

Ages: 13 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 110 (Actual)
Dates: Start 2013-02; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Number of study participants who chose long-acting reversible contraception (LARC) after all contraceptive counseling was done. | at enrollment/baseline visit
  This data was obtained by the number of participants who chose to have an IUD or Implant inserted after counseling at their clinic visit.

SECONDARY OUTCOMES:
Number of participants who maintained LARC uptake | 4 months from enrollment/baseline visit
  This data is being obtained through a brief follow-up questionnaire conducted over the phone.
Number of participants who maintained a positive opinion of LARC method as their primary choice for birth control | 4 months after enrollment/baseline visit.
  This data is being obtained through a brief follow-up questionnaire conducted over the phone.

CONTACTS AND LOCATIONS:
Overall Officials: Courtney A Schreiber, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States